CLINICAL TRIAL: NCT00345306
Title: Artificial Endometrial Preparation for Frozen Thawed Embryo Transfer Applying Either Endometrin or Utrogestan - a Clinical Comparative Study
Brief Title: Artificial Endometrial Preparation for Frozen Thawed Embryo Transfer Applying Either Endometrin or Utrogestan
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: no patient was recruited till 1/2008
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EndoUtro-HMO-CTIL
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2006-06

CONDITIONS: Frozen Thawed Embryo Transfer
Keywords: endometrial preparation; Utrogestan; Endometrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Comparison between two different progesterone administration

SUMMARY:
The transfer of frozen-thawed embryos can be performed in a natural ovulatory cycle or in a hormonally manipulated cycle with a comparable pregnancy rate of 15%-20% per ET. When a hormonally modulated ET cycle is scheduled,an artificial endometrial preparation is carried out using estrogen stimulation followed by a concomitant progesterone treatment. Two progestative drugs are currently used in conventional IVF treatment, Utrogetan and Endometrin. Although Endometrin has been be efficiently used to support the luteal phase after embryo transfer in IVF cycles, currently, there is no study that assess its efficacy for clinical use in frozen-thawed ET cycles. The present study aims to compare the outcome of frozen thawed ET cycles when either Endometrin or Utrogestan are used as the progestative substitution in an artificially prepared endometrium.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing frozen thawed ET cycles
2. Patient has at least two embryos suitable for transfer after thawing
3. Age 18-35 years -

Exclusion Criteria:

1. Any known sensitivity to Endometrin or Utrogestan
2. Endometrial thickness less than 7.5 mm after estrogen priming -

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Pregnancy rates

SECONDARY OUTCOMES:
Lutheal hormonal profile

CONTACTS AND LOCATIONS:
Overall Officials: Alex Simon, Principal Investigator — Hadassah University Hospital
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Simon Alex, Jerusalem